CLINICAL TRIAL: NCT04069754
Title: Passport to Freedom: Adaptation and Implementation of a Wellness Program to Educate and Empower Women Living in Transitional Housing Due to Intimate Partner Violence
Brief Title: Passport to Freedom (P2F): Adaptation and Implementation of a Wellness Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of staff to conduct study
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00203504
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Trauma
Keywords: trauma; stress; depression; coping; mindfulness
MeSH Terms: conditions — Wounds and Injuries; Depression

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention. There are no other groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Passport to Freedom Intervention Arm (Experimental): The intervention consists of 5 weekly, 90 minute group sessions that cover topics such as mindfulness, health, healthy relationships, family matters, and reflections
  Interventions: Behavioral: Adapted Passport to Freedom

INTERVENTIONS:
Behavioral: Adapted Passport to Freedom — 5 weekly, 90 minute group sessions that cover topics such as mindfulness, health, healthy relationships, family matters, and reflections.

SUMMARY:
Women currently residing at an emergency shelter for women and children will participate in group sessions that cover topics that promote physical and emotional well-being through a combination of mindfulness exercises and health promotion activities..

DETAILED DESCRIPTION:
In a group setting, the intervention will cover topics such as Mindfulness, Health (examine impact of trauma and stress on physical and mental well-being), Healthy relationships, Family matters (coping with conflicts) and Reflection session.

Each group session (5) will last approximately 90 minutes, once weekly, and begin and end with mindfulness exercises. The women are also encouraged to download free mindfulness apps to practice the exercises between sessions.

Women enrolled will receive health information that will cover a range of chronic health topics (pain, asthma, hypertension, diabetes, obesity), to complement already existing tools on mental health and post traumatic syndrome.

Women enrolled will complete surveys:

baseline questionnaires, a pre and post survey during each session, and follow-up questionnaires 4 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to read and write English
* Currently residing at the House of Ruth Maryland emergency shelter or onsite transitional housing.

Exclusion Criteria:

* Under 18 years of age
* Inability to speak or write English
* Physical or mental health conditions that would prevent meaningful group participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Change in Physical Health as assessed by the Perceived Health Competence Scale | Baseline, 9 weeks
  The Perceived Health Competence Scale measures the degree to which an individual feels capable of effectively managing their health. The score could range from 2-10. The higher the score, the greater the patient's perceived health competence.
Change in Mental Health as assessed by the Patient Health Questionnaire | Baseline, 9 weeks
  Patient Health Questionnaire assesses patient's level of distress and functional impairment. Score ranges from 0-4 depression severity is minimal or none. Score range from 5-9 is mild depression severity. Score range from 10-14 is moderate depression severity. 15-19 range is moderately severe depression. Range 20-27 indicates severe depression.

SECONDARY OUTCOMES:
Change in Stress as assessed by Everyday Stressor Index | Baseline, 9 weeks
  The Everyday Stressor Index assesses the problems faced on a daily basis by low-income mothers with young children. The instrument has a possible range of 20-80. A higher score indicates a higher level of daily stress.
Change in Emotions as assessed by Difficulties in Emotion Regulation Scale-Short Form | Baseline, 9 weeks
  The Difficulties in Emotion Regulation Scale is a self report measure of subjective emotion ability. The measure yields a total score sum as well as scores on six sub-scales. All subscales are scored so that higher values reflect greater difficulty with emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Patty Wilson, PhD, RN, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- House of Ruth Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.